CLINICAL TRIAL: NCT01324349
Title: A Prospective, Multi-Center, Randomized, Single-Blind Study to Compare the Hemostatic Patch to Fibrin Sealant (TachoSil®) in Subjects Undergoing Hepatic Surgery
Brief Title: Comparison of the Hemostatic Patch to Fibrin Sealant (TachoSil®) in Subjects Undergoing Hepatic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COVEULV0032
Record Dates: First submitted 2011-03-24; First posted 2011-03-29 (Estimated); Results first posted 2012-09-12 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-01

CONDITIONS: Liver Disease
Keywords: Hepatic; Topical Hemostat
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Veriset Hemostatic Patch (Experimental): Veriset Hemostatic Patch
  Interventions: Device: Veriset Hemostatic Patch
- Fibrin Sealant (TachoSil®) (Active Comparator): Fibrin Sealant (TachoSil®)
  Interventions: Device: Fibrin Sealant (TachoSil®)

INTERVENTIONS:
Device: Veriset Hemostatic Patch — Topical hemostat
  Arms: Veriset Hemostatic Patch
Device: Fibrin Sealant (TachoSil®) — Topical hemostat
  Arms: Fibrin Sealant (TachoSil®)

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of Covidien's Hemostatic Patch to control bleeding during hepatic surgery. The performance of the Hemostatic Patch will be compared to Control as an adjunct to conventional hemostatic techniques.

ELIGIBILITY:
Major Inclusion Criteria:

* Scheduled for non-emergent, hepatic surgery
* Presence of an appropriate target bleeding site (TBS) as defined by the protocol

Major Exclusion Criteria:

* Subject will be undergoing a laparoscopic hepatic procedure where the Hemostatic Patch will be delivered and applied through a trocar
* In subjects with documented history of cirrhosis, subject has uncorrected platelet count <60,000 per mm³ as determined by laboratory tests performed immediately prior to surgery
* Subject has severe coagulopathy defined as INR > 2.0
* Subject has Total Bilirubin >2.5mg/dL
* Subject has an active local infection at the Target Bleeding Site
* Study procedure involves a liver transplant recipient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-02; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Pollack, MD, Study Director — Medtronic - MITG
Locations (6):
- Innsbruck, Austria
- Belgium (2):
  - Ghent
  - Leuven
- Germany (3):
  - Hanover
  - Heidelberg
  - München

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who were scheduled for non-emergent, open hepatic surgery were assessed for potential study eligibility via a screening/baseline assessment performed within 30 days of their scheduled procedure.
Pre-assignment Details: Subjects who met the pre-operative eligibility criteria were considered for study participation. During the surgical procedures, subjects who met the intra-operative eligibility criteria were randomized. Subjects who did not meet all criteria were considered screen failures and not randomized.
Groups:
- Veriset Hemostatic Patch: Subject received the topical hemostat Veriset Hemostatic Patch
- Fibrin Sealant (TachoSil®): Subject received the topical hemostat TachoSil®
Period: Overall Study
Arm/Group | Veriset Hemostatic Patch | Fibrin Sealant (TachoSil®)
Started | 32 | 18
Completed | 31 | 16
Not Completed | 1 | 2
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Veriset Hemostatic Patch | Fibrin Sealant (TachoSil®) | Total
Number analyzed (Participants) | 32 | 18 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 12 | 26
  >=65 years | 18 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (14.9) | 62 (10.6) | 62.1 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 11 | 30
  Male | 13 | 7 | 20
Region of Enrollment [Number; unit: participants]
  Belgium | 11 | 5 | 16
  Austria | 6 | 4 | 10
  Germany | 15 | 9 | 24

OUTCOME MEASURES:

1. Primary Outcome: Median Time to Achieve Hemostasis Following Application of Study Treatment.
Description: Stopwatches will be provided to document time to hemostasis. Hemostasis will be assessed every 30 seconds until the 5-minute time point, at which point the visual inspection will continue at one-minute intervals up to 10 minutes or until hemostasis is achieved.
Time Frame: Intra-operative (day 1)
Population: Per the study protocol, the ITT population will serve as the primary analysis population for effectiveness. One randomized subject, Subject 1104, did not receive the assigned treatment (TachoSil®).
Measure: Median (Full Range); unit: Minutes
Arm/Group | Veriset Hemostatic Patch | Fibrin Sealant (TachoSil®)
Number analyzed (Participants) | 32 | 17
Minutes | 1 [0.5 to 4.0] | 3 [3 to 6.0]
Statistical Analysis 1: Comparison: Veriset Hemostatic Patch vs Fibrin Sealant (TachoSil®); The primary effectiveness endpoint was time to hemostasis. The Kaplan-Meier method was used to estimate the survival distribution and to obtain the estimated median time to hemostasis for each treatment. Subjects who did not achieve hemostasis by 10 minutes were to be censored as of that time point. For each treatment, 95% Brookmeyer-Crowley confidence intervals for the median were computed based upon the sign test; Test type: Superiority or Other; p < 0.0001, Log Rank; Median Difference (Final Values) = 2 — Median difference equals control median minus Hemostatic Patch median in minutes

2. Secondary Outcome: Number of Subjects to Achieve Hemostasis Within 3 Minutes of Study Treatment Application
Description: as for outcome 1
Time Frame: Intra-operative (day 1)
Population: Per the study protocol, the ITT population will serve as the primary analysis population for effectiveness and will be discussed in this report. One randomized subject, Subject 1104, did not receive the assigned treatment (TachoSil).
Measure: Number; unit: Participants
Arm/Group | Veriset Hemostatic Patch | Fibrin Sealant (TachoSil®)
Number analyzed (Participants) | 32 | 17
Participants | 30 [77.8 to 98.9] | 12 [46.0 to 88.0]
Statistical Analysis 1: Comparison: Veriset Hemostatic Patch vs Fibrin Sealant (TachoSil®); The secondary effectiveness endpoint was hemostasis within 3 minutes. The number and percentage of subjects who achieved hemostasis within 3 minutes are presented for each treatment group. The proportions of subjects who achieved hemostasis within 3 minutes were compared between treatments using the Suissa and Shuster test. Additionally, a 95% Blyth-Still-Casella confidence interval for the true proportion was computed for each treatment; Test type: Superiority or Other; p = 0.0339, Suissa and Shuster test; Risk Difference (RD) = 23.2, 95% CI 2-sided [1.9 to 47.3] — Risk difference equals percentage hemostasis for Hemostatic Patch minus percentage hemostasis for control

3. Secondary Outcome: Number of Subjects With Treatment-emergent Adverse Events
Time Frame: Up to 30 days post surgery.
Population: All treated subjects are included in the Safety population.
Measure: Number; unit: Participants
Arm/Group | Veriset Hemostatic Patch | Fibrin Sealant (TachoSil®)
Number analyzed (Participants) | 32 | 17
Participants | 23 | 14
Statistical Analysis 1: Comparison: Veriset Hemostatic Patch vs Fibrin Sealant (TachoSil®); The incidence of subjects experiencing treatment-emergent adverse events (TEAEs) (defined under this protocol as Adverse Events) was summarized by MedDRA system organ class (SOC) and preferred term (PT) for each treatment group for the safety population. Tests for differences between the two treatments in the proportion of subjects experiencing any adverse event were made using Fisher's Exact Test; Test type: Superiority or Other; p = 0.5029, Fisher Exact; Risk Difference (RD) = 10.5 — Risk difference equals percent of subjects with any treatment emergent adverse events in control group minus percent of subjects with any treatment emergent adverse events in Hemostatic Patch group

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of randomization through the 30 day follow-up visit.
Arm/Group | Veriset Hemostatic Patch | Fibrin Sealant (TachoSil®)
Serious Adverse Events (participants affected / at risk) | 10/32 | 8/17
Other Adverse Events (participants affected / at risk) | 22/32 | 10/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Veriset Hemostatic Patch (N=32) | Fibrin Sealant (TachoSil®) (N=17)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 1 (1)
Biloma (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 1 (1)
Haematoma infection (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 2 (2)
Pyothorax (Infections and infestations) | 0 (0) | 1 (1)
Post procedural bile leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Inferior vena caval occlusion (Vascular disorders) | 1 (1) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Veriset Hemostatic Patch (N=32) | Fibrin Sealant (TachoSil®) (N=17)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal compartment syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 5 (6) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Papilla of Vater stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Inflammation (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 2 (2)
Biloma (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 4 (4) | 1 (1)
Bacterial infection (Infections and infestations) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Weaning failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Metastases to chest wall (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to diaphragm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure actute (Renal and urinary disorders) | 1 (1) | 1 (1)
Urge incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No